CLINICAL TRIAL: NCT05876910
Title: Neural Mechanisms for Stopping Ongoing Speech Production
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K99DC020235 (NIH); K99DC020235 (NIH)
Record Dates: First submitted 2023-05-11; First posted 2023-05-26 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Epilepsy; Speech
MeSH Terms: conditions — Epilepsy; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voice and Electrocorticography (ECoG) recording during Speech Production Tasks (Experimental): Participants produce speech following visual cues on a computer while ECoG signals for neural activity and voice was recorded during their inpatient hospitalization at the University of California, San Francisco (UCSF).
  Interventions: Behavioral: Speech Production Tasks

INTERVENTIONS:
Behavioral: Speech Production Tasks — View visual cues and undergo speech production for 30 minutes. Electrical stimulation of speech related brain regions in the middle of speech production.

SUMMARY:
Speech and communication disorders often result in aberrant control of the timing of speech production, such as making improper stops at places where they should not be. During normal speech, the ability to stop when necessary is important for maintaining turn-taking in a smooth conversation. Existing studies have largely investigated neural circuits that support the preparation and generation of speech sounds. It is believed that activity in the prefrontal and premotor cortical areas facilitates high-level speech control and activity in the ventral part of the sensorimotor cortex controls the articulator (e.g. lip, jaw, tongue) movements. However, little is known about the neural mechanism controlling a sudden and voluntary stop of speech. Traditional view attributes this to a disengagement of motor signals while recent evidence suggested there may be an inhibitory control mechanism. This gap in knowledge limits our understanding of disorders like stuttering and aphasia, where deficits in speech timing control are among the common symptoms. The overall goal of this study is to determine how the brain controls the stopping of ongoing speech production to deepen our understanding of speech and communication in normal and impaired conditions.

DETAILED DESCRIPTION:
High-density electrocorticography (ECoG) is a state-of-the-art technique with fine spatial and temporal resolutions that are well suited for studying the neural dynamics of speech. This study proposes to assess speech production in patients who are undergoing high-density ECoG recording to carry out clinical procedures for indications related to their medical condition. The research study team will investigate neural signals correlated with speech stopping using speech production and stopping tasks with visual cues. Electrical stimulation routinely used for language mapping will also be applied to test the causal effect on speech behavior in brain areas found to be activated during the speech tasks. The research study team will compare effects on neural activity and behavior within each individual subject and identify common patterns of activity across subjects. The aims of this study seek to define the premotor signal for the control of speech stopping (Aim 1), determine the effect of stop activity on articulatory control during stopping (Aim 2), and determine the role of the premotor network for stopping in conversation contexts (Aim 3). These aims will provide basic knowledge for the precise control of speech stopping and the control of speech timing in general, bridging the current speech production studies to real-world communication conditions, and help inspire new theories of speech motor control.

ELIGIBILITY:
Inclusion Criteria:

* Participants with medication refractory epilepsy at UCSF undergoing surgical electrode implantation of subdural electrode arrays to define their seizure focus and
* Participants with electrodes implanted who are willing and able to cooperate with study tasks.

Exclusion Criteria:

* Participants who lack capacity,
* Participants who decline to provide informed consent or
* Participants with cognitive deficits that preclude reliable completion of study tasks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12-08 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Neural Activity | During inpatient hospitalization, up to 14 days after surgical electrode implantation
  The mean change in neural activity is calculated as the average change in neural activity across trials between a time period (~1 second) after the visual cue and a time period (~1 second) before the visual cue. Included neural activity is within the 30-minute period of cue viewing and speech production tasks.

SECONDARY OUTCOMES:
Number of sites with stimulation induced speech termination | During inpatient hospitalization, up to 14 days after surgical electrode implantation
  The sites with stimulation induced speech termination are defined as the stimulation sites where termination of speech production (occurrence) is observed within 10 seconds after the electrical stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Lingyun Zhao, PhD, Principal Investigator — University of California, San Francisco; Edward F Chang, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No